CLINICAL TRIAL: NCT00564785
Title: A Randomized, Double-Blind, Controlled Trial of the Synera™ vs. Lidocaine for Epidural Needle Insertion in Laboring Women
Brief Title: Synera™ for Epidural Needle Insertion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: IWK Health Centre (Other)
Collaborators: Duke University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DWA-2007-001
Record Dates: First submitted 2007-11-27; First posted 2007-11-28 (Estimated); Last update posted 2007-11-28 (Estimated); Status verified 2007-01

CONDITIONS: Pain Associated With Epidural Needle Insertion

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo patch
- Synera(TM) (Experimental)
  Interventions: Drug: Synera(TM)

INTERVENTIONS:
Drug: Synera(TM) — Synera(TM) patch applied 20 minutes prior to epidural
  Arms: Synera(TM)
Other: Placebo patch — placebo patch applied 20 minutes prior to epidural
  Arms: Placebo

SUMMARY:
We hypothesized that the analgesic effect of Synera™ analgesic patch would be superior to traditional infiltration with lidocaine for pain of epidural needle insertion in laboring parturients.

ELIGIBILITY:
Inclusion Criteria:

* older than 18 years, body mass index less than 45 kg•m-2, requesting a labor epidural

Exclusion Criteria:

* hypersensitivity to any study medications

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2007-02; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Subject VRS (0 - 11) with epidural needle insertion | 1 hour

SECONDARY OUTCOMES:
Anesthesia provider perceived VRS | 1 hour
Need for deep infiltration with local anesthesia | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Ronald B George, MD FRCPC, Principal Investigator — IWK Health Centre
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States